CLINICAL TRIAL: NCT03385876
Title: Rapid Whole Genome Sequencing (rWGS): Rapid Genomic Sequencing for Acutely Ill Patients and the Collection, Storage, Analysis, and Distribution of Biological Samples, Genomic and Clinical Data
Brief Title: Rapid Whole Genome Sequencing Study
Acronym: rWGS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Responsible Party: Principal Investigator, David Dimmock, MD, Medical Director, Rady Pediatric Genomics & Systems Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rWGS Protocol #20171726
Record Dates: First submitted 2017-12-13; First posted 2017-12-29 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Genetic Diseases; Genetic Syndrome
Keywords: Rady Children's; Pediatric; Genomic; Precision Medicine; Biorepository
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrollees (Experimental): Enrollment of healthy and affected subjects to collect samples and data for a pediatric genomic biorepository. Data includes genomic sequencing and resultant molecular diagnostic results, if any.
  Interventions: Genetic: Genomic sequencing and molecular diagnostic results, if any

INTERVENTIONS:
Genetic: Genomic sequencing and molecular diagnostic results, if any — Samples will be stored in the pediatric genomic biorepository. A subset of samples will undergo genetic/genomic analysis.
  Other Names: Pediatric Genetic Biorepository; Pediatric Precision Medicine

SUMMARY:
Rapid Whole Genome Sequencing (rWGS) has proven to provide much faster diagnoses than traditional clinical testing, including clinical Whole Exome Sequencing (WES) and standard Whole Genome Sequencing (WGS). This collaborative study seeks to provide rWGS as a research test to additional pediatric hospitals nationwide to assist in the rapid diagnosis of acutely ill children suspected of a genetic condition. The study will examine diagnosis rates, changes in clinical care as a result of a genetic diagnosis, and health economics including potential cost-effectiveness of rWGS. This study will also serve as a biorepository for future research on samples and data generated from genomic sequencing.

DETAILED DESCRIPTION:
Rapid Whole Genome Sequencing (rWGS) is a new technology that is able to deliver symptom-driven diagnoses of childhood-onset genetic diseases in as little as 26 hours. Investigators at RCIGM have shown that rWGS has higher diagnostic rates than traditional molecular testing in acutely ill infants suspected of a genetic diagnosis, with diagnostic rates up to 57%. Similarly, in the infant population, RCIGM researchers have shown that these diagnoses are useful in directing clinical care, with up to 70% of infants who receive a diagnosis having a subsequent change in management. In some cases, a timely diagnosis results in treatments that are lifesaving. RCIGM investigators have shown that up to 25% of infants who receive a diagnosis have a subsequent change in management that prevents morbidity. More data is needed to determine whether these results are found at other institutions, among other ethnic and racial groups, and in larger numbers of patients. More data is needed to examine the acute and long-term clinical utility of such testing, both in newborns and older children, as well as to determine the cost-effectiveness of this testing for other institutions. As such, this study will be a collaboration of multiple sites to share data and experiences of rWGS with the scientific community as well as hospital administrations, insurance companies and other key stakeholders who may be interested in promoting rWGS as a first-line clinical test in the future.

The study will provide clinical laboratory-confirmed results related to the affected patient's symptoms, including optional incidental findings unless subjects opt-out for these additional results, to allow for these research findings to be used in clinical care. Furthermore, this study will aggregate data regarding standard clinical genetic testing from multiple sites as well as cost measures to not only identify differences in diagnostic rates, diagnostic accuracy, and times to diagnoses, but to determine the cost-effectiveness of this testing and subsequent changes in care management. Clinical utility will be defined as changes in care that follow directly from results of genetic testing (both positive and negative), including standard clinical tests and rWGS. This data will be used to further examine the analytic, diagnostic, and clinical utility and cost-effectiveness of this testing.

rWGS methods continue to improve, and pediatric genomic medicine is a very new field of medical practice. This study will also inform investigators regarding best practices, both in terms of traditional medical outcomes and patient-centered outcomes. Consequently, this study will also act as a biorepository for samples and data as the ability to share genomic and phenotypic data amongst researchers is critical to progressing our understanding of the nascent field of pediatric genomic medicine.

Specific Aims:

1. To collect biological samples and associated clinical data from acutely ill pediatric patients who may have a genetic disease and their family members (Phenome).
2. To create, analyze and store genomic data from the biological samples. Genomic data will include genomic (gDNA) sequences, RNA sequences, and/or other related 'omic data (including, but not limited to, pharmacogenomics, transcriptomics, and epigenomics). Genomic data from rWGS will include single nucleotide calls (SNVs), structural variants such as copy number testing, genomic rearrangements, gene expression , the "whole transcriptome" or more limited DNA sequencing panels of specific genes or of all exons of genes (the "Exome").
3. To evaluate the diagnosis rate of genetic diseases by rWGS in an acutely ill population enrolling from multiple sites with comparisons to standard clinical genetic testing.
4. To assess the clinical utility of rapid genetic diagnoses in the care and management of patients.
5. To examine the health economics and cost-effectiveness of this rapid testing across many sites.
6. To investigate and improve genomics technologies and software to enhance understanding and testing abilities related to childhood diseases and potential treatment responses.
7. To make specimens and data available for qualified researchers and collaborators to further the understanding of rare childhood diseases and treatment responses.
8. To collect and correlate genomic data from a wide variety of populations and clinical presentations.
9. To provide sample and data collections with uniform consent, methods of acquisition, storage for genome-based research studies with subsequent IRB approvals.
10. To analyze and report clinically-confirmed genomic diagnoses and treatment guidance through use of new research technologies.
11. To identify and study novel gene and disease processes.

ELIGIBILITY:
Inclusion Criteria:

* The Repository will be comprised of samples from symptomatic patients, individuals reported to be their (symptomatic or asymptomatic) biologic family members, and control individuals. In this context a "symptomatic patient" is characterized as a patient whose treating physician has identified phenotypic features and/or signs of illness potentially attributable to a genetic disorder (also referred to as "Affected" or "Proband"). There will be no age, gender, race, or health restrictions for this Biorepository Study. However, since this study will be performed at children's hospitals and since genetic disorders are more likely to be present in children less than 4 months of age these cases will likely be preferentially enrolled. Preference will also be given to those who are acutely ill, suspected of a genetic condition, and for whom a diagnosis may result in change of clinical management.

Exclusion Criteria:

* Participants will be excluded if they are unwilling to consent to research.

A patient may be determined ineligible if there is a prior diagnosis that explains their clinical presentation, if other traditional clinical genetic testing is more appropriate at the time of referral, if the clinical presentation is insufficient at the time of referral to suggest a genetic etiology, if the parents are unable or unwilling to provide permission for participation, if child protective services is involved in the case unless the child's life is in immediate danger and research holds out a prospect of direct benefit that is important to the health or well-being of the child and is available only in the context of the research in which case permission will be obtained from the party legally responsible for medical decisions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of samples enrolled per year | Yearly through study completion estimated to be 40 years.
  Establishment of a biorepository for genomic/precision medicine use in pediatric population. This will make samples available to study rare genetic disorders, screening methods, diagnostic methods, other "omics," and bench research for possible treatments.

SECONDARY OUTCOMES:
Proportion of children receiving molecular diagnoses | Through study completion estimated to be 40 years.
  Utilize cutting edge technologies to improve both diagnostic rates and time to diagnosis for rare genetic diseases. Symptom driven return of results and analysis of clinical utility.
Time taken to receive molecular diagnosis | From date of enrollment until the date of documented clinical laboratory diagnosis or date of death from any cause, whichever came first, assessed up to 10 years.
Proportion of children in which human phenotype ontology (HPO) terms accurately predict molecular diagnosis | Through study completion estimated to be 40 years.
Subject's main provider's perceived clinical utility of genomic sequencing | Within one month of the return of results.
  Perceived utility/benefit of sequencing based on "Clinician Assessment" scale completed by patient's providers.
Comparing diagnostic rates between singleton and trio analysis | Within 30 days of enrollment.
  Marginal increase in diagnostic yield above singleton analysis based on the number of clinically confirmed diagnoses posted in medical record following singleton and trio levels of analysis in cases when both biological parents are available.

CONTACTS AND LOCATIONS:
Overall Officials: David Dimmock, MD, Principal Investigator — Rady Pediatric Genomics & Systems Medicine Institute; Stephen Kingsmore, Study Director — Rady Pediatric Genomics & Systems Medicine Institute
Locations (1):
- Rady Children's Institute for Genomic Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Owen MJ, Niemi AK, Dimmock DP, Speziale M, Nespeca M, Chau KK, Van Der Kraan L, Wright MS, Hansen C, Veeraraghavan N, Ding Y, Lenberg J, Chowdhury S, Hobbs CA, Batalov S, Zhu Z, Nahas SA, Gilmer S, Knight G, Lefebvre S, Reynders J, Defay T, Weir J, Thomson VS, Fraser L, Lajoie BR, McPhail TK, Mehtalia SS, Kunard CM, Hall KP, Kingsmore SF. Rapid Sequencing-Based Diagnosis of Thiamine Metabolism Dysfunction Syndrome. N Engl J Med. 2021 Jun 3;384(22):2159-2161. doi: 10.1056/NEJMc2100365. No abstract available. PMID 34077649
- [Result] Friedman J, Bird LM, Haas R, Robbins SL, Nahas SA, Dimmock DP, Yousefzadeh MJ, Witt MA, Niedernhofer LJ, Chowdhury S. Ending a diagnostic odyssey: Moving from exome to genome to identify cockayne syndrome. Mol Genet Genomic Med. 2021 Jul;9(7):e1623. doi: 10.1002/mgg3.1623. Epub 2021 Jun 2. PMID 34076366
- [Result] Rossignol F, Duarte Moreno MS, Benoist JF, Boehm M, Bourrat E, Cano A, Chabrol B, Cosson C, Diaz JLD, D'Harlingue A, Dimmock D, Freeman AF, Garcia MT, Garganta C, Goerge T, Halbach SS, de Laffolie J, Lam CT, Martin L, Martins E, Meinhardt A, Melki I, Ombrello AK, Perez N, Quelhas D, Scott A, Slavotinek AM, Soares AR, Stein SL, Sussmuth K, Thies J, Ferreira CR, Schiff M. Quantitative analysis of the natural history of prolidase deficiency: description of 17 families and systematic review of published cases. Genet Med. 2021 Sep;23(9):1604-1615. doi: 10.1038/s41436-021-01200-2. Epub 2021 May 26. PMID 34040193
- [Result] Sweeney NM, Nahas SA, Chowdhury S, Batalov S, Clark M, Caylor S, Cakici J, Nigro JJ, Ding Y, Veeraraghavan N, Hobbs C, Dimmock D, Kingsmore SF. Rapid whole genome sequencing impacts care and resource utilization in infants with congenital heart disease. NPJ Genom Med. 2021 Apr 22;6(1):29. doi: 10.1038/s41525-021-00192-x. PMID 33888711
- [Result] Kuehn HS, Gloude NJ, Dimmock D, Tokita M, Wright M, Rosenzweig SD, Collins C. Abnormal SCID Newborn Screening and Spontaneous Recovery Associated with a Novel Haploinsufficiency IKZF1 Mutation. J Clin Immunol. 2021 Aug;41(6):1241-1249. doi: 10.1007/s10875-021-01035-1. Epub 2021 Apr 14. PMID 33855675
- [Result] Rusert JM, Juarez EF, Brabetz S, Jensen J, Garancher A, Chau LQ, Tacheva-Grigorova SK, Wahab S, Udaka YT, Finlay D, Seker-Cin H, Reardon B, Grobner S, Serrano J, Ecker J, Qi L, Kogiso M, Du Y, Baxter PA, Henderson JJ, Berens ME, Vuori K, Milde T, Cho YJ, Li XN, Olson JM, Reyes I, Snuderl M, Wong TC, Dimmock DP, Nahas SA, Malicki D, Crawford JR, Levy ML, Van Allen EM, Pfister SM, Tamayo P, Kool M, Mesirov JP, Wechsler-Reya RJ. Functional Precision Medicine Identifies New Therapeutic Candidates for Medulloblastoma. Cancer Res. 2020 Dec 1;80(23):5393-5407. doi: 10.1158/0008-5472.CAN-20-1655. Epub 2020 Oct 12. PMID 33046443
- [Result] Ramchandar N, Ding Y, Farnaes L, Dimmock D, Hobbs C, Kingsmore SF, Bainbridge M. Diagnosis of cytomegalovirus infection from clinical whole genome sequencing. Sci Rep. 2020 Jul 3;10(1):11020. doi: 10.1038/s41598-020-67656-5. PMID 32620939
- [Result] Chandrasekar I, Tourney A, Loo K, Carmichael J, James K, Ellsworth KA, Dimmock D, Joseph M. Hemimegalencephaly and intractable seizures associated with the NPRL3 gene variant in a newborn: A case report. Am J Med Genet A. 2021 Jul;185(7):2126-2130. doi: 10.1002/ajmg.a.62185. Epub 2021 Mar 22. PMID 33749980
- [Result] Tokita MJ, Nahas S, Briggs B, Malicki DM, Mesirov JP, Reyes IAC, Farnaes L, Levy ML, Kingsmore SF, Dimmock D, Crawford JR, Wechsler-Reya RJ. Biallelic loss of GNAS in a patient with pediatric medulloblastoma. Cold Spring Harb Mol Case Stud. 2019 Oct 23;5(5):a004572. doi: 10.1101/mcs.a004572. Print 2019 Oct. PMID 31624069
- [Result] Kadakia S, Farnaes L, Dimmock D, Chowdhury S, Ding Y, Anderson EJ, Kingsmore S, Newfield RS. Diagnosis and treatment of a boy with IPEX syndrome presenting with diabetes in early infancy. Clin Case Rep. 2019 Sep 27;7(11):2123-2127. doi: 10.1002/ccr3.2438. eCollection 2019 Nov. PMID 31788263
- [Result] Clark MM, Hildreth A, Batalov S, Ding Y, Chowdhury S, Watkins K, Ellsworth K, Camp B, Kint CI, Yacoubian C, Farnaes L, Bainbridge MN, Beebe C, Braun JJA, Bray M, Carroll J, Cakici JA, Caylor SA, Clarke C, Creed MP, Friedman J, Frith A, Gain R, Gaughran M, George S, Gilmer S, Gleeson J, Gore J, Grunenwald H, Hovey RL, Janes ML, Lin K, McDonagh PD, McBride K, Mulrooney P, Nahas S, Oh D, Oriol A, Puckett L, Rady Z, Reese MG, Ryu J, Salz L, Sanford E, Stewart L, Sweeney N, Tokita M, Van Der Kraan L, White S, Wigby K, Williams B, Wong T, Wright MS, Yamada C, Schols P, Reynders J, Hall K, Dimmock D, Veeraraghavan N, Defay T, Kingsmore SF. Diagnosis of genetic diseases in seriously ill children by rapid whole-genome sequencing and automated phenotyping and interpretation. Sci Transl Med. 2019 Apr 24;11(489):eaat6177. doi: 10.1126/scitranslmed.aat6177. PMID 31019026
- [Result] Kingsmore SF, Ramchandar N, James K, Niemi AK, Feigenbaum A, Ding Y, Benson W, Hobbs C, Nahas S, Chowdhury S, Dimmock D. Mortality in a neonate with molybdenum cofactor deficiency illustrates the need for a comprehensive rapid precision medicine system. Cold Spring Harb Mol Case Stud. 2020 Feb 3;6(1):a004705. doi: 10.1101/mcs.a004705. Print 2020 Feb. PMID 32014857
- [Result] Friedman J, Smith DE, Issa MY, Stanley V, Wang R, Mendes MI, Wright MS, Wigby K, Hildreth A, Crawford JR, Koehler AE, Chowdhury S, Nahas S, Zhai L, Xu Z, Lo WS, James KN, Musaev D, Accogli A, Guerrero K, Tran LT, Omar TEI, Ben-Omran T, Dimmock D, Kingsmore SF, Salomons GS, Zaki MS, Bernard G, Gleeson JG. Biallelic mutations in valyl-tRNA synthetase gene VARS are associated with a progressive neurodevelopmental epileptic encephalopathy. Nat Commun. 2019 Feb 12;10(1):707. doi: 10.1038/s41467-018-07067-3. PMID 30755602